CLINICAL TRIAL: NCT02932046
Title: Hunger and Satiety Perception in Patients With Anorexia Nervosa
Brief Title: Hunger and Satiety in Anorexia Nervosa
Acronym: HUSAAN
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, René Klinkby Støving, Chief physician, Associate Professor, PhD., Odense University Hospital
Other Study IDs: HUSAAN
Record Dates: First submitted 2016-07-05; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-07

CONDITIONS: Anorexia Nervosa; Appetite Disorders
Keywords: eating disorders; anorexia nervosa; appetite
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standardized noon meal: Patients with anorexia nervosa during in-patient treatment are rating hunger and satiety on a visual analogue scale before and after a standardized and supervised meal. The meal is "treatment as usual" in a specialized ward. A patient may participate several times, if readmitted.
  Interventions: Dietary Supplement: Standardized noon meal

INTERVENTIONS:
Dietary Supplement: Standardized noon meal — The meal is "treatment as usual" in the specialized somatic stabilization ward for patients with severe anorexia nervosa.

SUMMARY:
Anorexia means loss of appetite. But there is disagreement about whether the appetite is changed by the disease anorexia nervosa (AN). Appetite is a subjective essential sense, which is regulated in a complex ensemble between brain, stomach - intestinal system and hormones. As a direct result of malnutrition, there are many somatic complications caused by the disease AN. Several of these complications may in itself affect hunger- and satiety perception. An example of this is delayed gastric emptying. Furthermore, changes in the hormone systems affects the biological "reward system" in the brain, which plays an important role in appetite regulation. There is clearly need for research that could lead to better treatments for AN. Hunger- and satiety perception has only been studied in a few small cross-sectional studies with no clear conclusion.

The purpose of the study is to determine whether a visual analog scale measurement can detect changes in hunger- and satiety perception in a least 30 patients admitted to nutrition for life-threatening severe anorexia nervosa. It may lead to the first step in the development of a simple and inexpensive instrument which may prove to be useful in measuring the impact of new and ongoing treatments of the disease.

DETAILED DESCRIPTION:
Appetite refers to the desire associated with eating. Both internal and external factors can stimulate appetite. Hunger and satiety are included in appetite regulation. Hunger is related to physiological needs and the commencement of eating. Satiety refers to a state without the urge to eat, where both the onset of satiety and post ingestion satiety are included.

Anorexia is abnormal loss of appetite for food. Anorexia nervosa is an eating disorder characterized by food restriction, despite low weight, leading to speculation about the presence of appetite alterations by weight loss.

AN is a syndrome of unknown etiology which has been well described since 1873, and which occurs most frequently in adolescent women. The syndrome is characterized by distorted body image, and fear of obesity, why low ideal weight is pursued. The disorder occurs in different degrees of severity with secondary endocrine and metabolic changes and disturbances. The symptoms may also include excessive physical activity, abuse of laxatives, or diuretics and self-induced vomiting.

There are multiple medical complications due to the starvation and weight loss in AN, several of which directly may affect appetite, for instance, delayed emptying of the stomach and constipation. Furthermore, compression of duodenum has been observed causing nausea and early satiety.

Hypothalamic hypogonadism is one of the well-known adaptive endocrine alterations in AN due to starvation and exaggerated exercise. Progesterone and testosterone is believed to stimulate appetite and eating, in a manner mediated centrally, selectively increasing the number of meals.

Moreover, AN patients have significantly higher levels of ghrelin, growth hormone (GH) and cortisol and significantly lower leptin, compared with partially recovered AN patients and constitutionally thin subjects.

Hunger and satiety are subjective sensations which may be influenced by sensory factors and palatability, including taste, smell and texture. A recent study suggested that patients with AN may have an altered perception of olfactory, gustatory stimuli, and reduced perception of bitter stimuli.

Other physiological factors such as, hypothalamic and mesolimbic endocannabinoids, enhance appetite by stimulating neurochemical pathways underlying both homeostatic and rewarding aspects of food intake. Endocannabinoids are involved in food-related reward mechanisms, and there are increasing evidence that these mechanisms are dysregulated in AN patients. Moreover, functional neuroimaging studies have demonstrated decreased food-related stimuli in brain areas of the mesolimbic reward system in AN patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe AN admitted to the specialized nutrition unit at Center for Eating disorders at Odense University Hospital are included.

Exclusion Criteria:

* Patients admitted only for short-term water-electrolyte correction, are excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with anorexia nervosa.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Hunger and satiety sensation | 30 minutes
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: René Stoving, PhD, Study Chair — Odense UH, Denmark
Locations (1):
- Center for eating Disorders, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gull WW. Anorexia nervosa (apepsia hysterica, anorexia hysterica). 1868. Obes Res. 1997 Sep;5(5):498-502. doi: 10.1002/j.1550-8528.1997.tb00677.x. No abstract available. PMID 9385628
- [Background] Stoving RK, Hangaard J, Hagen C. Update on endocrine disturbances in anorexia nervosa. J Pediatr Endocrinol Metab. 2001 May;14(5):459-80. doi: 10.1515/jpem.2001.14.5.459. PMID 11393567
- [Background] Westmoreland P, Krantz MJ, Mehler PS. Medical Complications of Anorexia Nervosa and Bulimia. Am J Med. 2016 Jan;129(1):30-7. doi: 10.1016/j.amjmed.2015.06.031. Epub 2015 Jul 10. PMID 26169883
- [Background] Asarian L, Geary N. Sex differences in the physiology of eating. Am J Physiol Regul Integr Comp Physiol. 2013 Dec;305(11):R1215-67. doi: 10.1152/ajpregu.00446.2012. Epub 2013 Jul 31. PMID 23904103
- [Background] Miljic D, Pekic S, Djurovic M, Doknic M, Milic N, Casanueva FF, Ghatei M, Popovic V. Ghrelin has partial or no effect on appetite, growth hormone, prolactin, and cortisol release in patients with anorexia nervosa. J Clin Endocrinol Metab. 2006 Apr;91(4):1491-5. doi: 10.1210/jc.2005-2304. Epub 2006 Jan 31. PMID 16449333
- [Background] Dazzi F, Nitto SD, Zambetti G, Loriedo C, Ciofalo A. Alterations of the olfactory-gustatory functions in patients with eating disorders. Eur Eat Disord Rev. 2013 Sep;21(5):382-5. doi: 10.1002/erv.2238. Epub 2013 Jun 20. PMID 23788398
- [Background] Stoving RK, Andries A, Brixen K, Flyvbjerg A, Horder K, Frystyk J. Leptin, ghrelin, and endocannabinoids: potential therapeutic targets in anorexia nervosa. J Psychiatr Res. 2009 Apr;43(7):671-9. doi: 10.1016/j.jpsychires.2008.09.007. Epub 2008 Oct 15. PMID 18926548
- [Background] Monteleone AM, Di Marzo V, Aveta T, Piscitelli F, Dalle Grave R, Scognamiglio P, El Ghoch M, Calugi S, Monteleone P, Maj M. Deranged endocannabinoid responses to hedonic eating in underweight and recently weight-restored patients with anorexia nervosa. Am J Clin Nutr. 2015 Feb;101(2):262-9. doi: 10.3945/ajcn.114.096164. Epub 2014 Dec 10. PMID 25646322
- [Background] Doucet E, Imbeault P, St-Pierre S, Almeras N, Mauriege P, Richard D, Tremblay A. Appetite after weight loss by energy restriction and a low-fat diet-exercise follow-up. Int J Obes Relat Metab Disord. 2000 Jul;24(7):906-14. doi: 10.1038/sj.ijo.0801251. PMID 10918539
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749